CLINICAL TRIAL: NCT06997627
Title: An Open(Part 1), Single-arm(Part 1), Randomized(Part 2), Double-blind(Part 2), Active-controlled(Part 2) Phase I/II Clinical Trial to Evaluate the Safety and Efficacy (Immunogenicity) of GC3111B in Healthy Adults
Brief Title: A Phase I/II Study to Evaluate the Safety and Immunogenicity of GC3111B in Healthy Adults
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GC Biopharma Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GC3111B_Tdap_P1201
Record Dates: First submitted 2025-05-15; First posted 2025-05-30 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Tetanus-diphtheria-acellular Pertussis (Tdap)
MeSH Terms: interventions — Boostrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC3111B (Experimental): Participants randomized to receive a single dose of GC3111B vaccine.
  Interventions: Biological: GC3111B
- Boostrix® (Active Comparator): Participants randomized to receive a single dose of Boostrix® vaccine.
  Interventions: Biological: Boostrix®

INTERVENTIONS:
Biological: GC3111B — 0.5 mL, Intramuscular injection
  Arms: GC3111B
Biological: Boostrix® — 0.5 mL, Intramuscular injection
  Arms: Boostrix®

SUMMARY:
This clinical trial consists of two parts: Part 1, which explores safety, and Part 2, which examines both safety and efficacy (immunogenicity). Part 1 is a single-center, open-label, single-group study, while Part 2 is designed as a multicenter, double-blind, randomized, active-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 to 64 years old as of the date of written consent.
* Individuals with no history of vaccination with a vaccine containing diphtheria, tetanus, or pertussis antigens within the past 2 years prior to administration of the investigational product.

Exclusion Criteria:

* Individuals who have received a vaccine within 4 weeks prior to administration of the investigational product.
* Individuals with a history of Tdap vaccination prior to administration of the investigational product.
* Pregnant and breastfeeding women.
* Individuals who have participated in other clinical trials involving investigational products/devices within 6 months prior to administration of the investigational product.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Solicited adverse events occurring by day 14 after administration of the investigational product | 14 days after administration of the IP
Unsolicited adverse events occurring by day 28 after administration of the investigational product | 28 days after administration of the IP
Acute adverse events occurring within 30 minutes after administration of the investigational product | 30 minutes after administration of the IP
Serious adverse events (SAE) and adverse events of special interest (AESI) occurring up to 180 days after administration of the investigational product | 180 days after administration of the IP
Clinically significant findings in vital signs, laboratory tests, 12-lead electrocardiograms, and physical examinations | 28 days after administration of the IP

SECONDARY OUTCOMES:
Antibody rates for diphtheria and tetanus on day 28 after administration of the investigational product | 28 days after administration of the IP
Boosting response rates for diphtheria, tetanus, and pertussis on day 28 after administration of the investigational product | 28 days after administration of the IP
  Boosting response rate: 1) If less than 0.1 IU/ml before vaccination, it should be 0.4 IU/ml or higher after the vaccination, or 2) if not less than 0.1 IU/ml before vaccination, it should be 4 times or higher after the vaccination.
Geometric mean concentrations (GMC) of antibodies against diphtheria, tetanus, and pertussis antitoxins (anti-PT, anti-FHA, anti-PRN) on day 28 after administration of the investigational product | 28 days after administration of the IP

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic Univ. of Korea Eunpyeong St. Mary's Hospital, Seoul, South Korea